CLINICAL TRIAL: NCT00794339
Title: Copper Cu 64-ATSM and PET/CT Scan in Predicting Disease Progression in Patients With Newly-Diagnosed Stage IB, Stage II, Stage III, or Stage IVA Cervical Cancer Who Are Undergoing Chemoradiotherapy Per NCCN Guidelines
Brief Title: Phase II Trial of 64Cu-ATSM PET/CT in Cervical Cancer
Acronym: ACRIN6682
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: transfer of funding
Sponsor: American College of Radiology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); American College of Radiology Imaging Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000624407; ACRIN-6682 (Other Grant/Funding Number: ACRIN Foundation); U01CA080098 (NIH); U01CA079778 (NIH)
Record Dates: First submitted 2008-11-19; First posted 2008-11-20 (Estimated); Results first posted 2021-01-28 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cervical Cancer
Keywords: cervical squamous cell carcinoma; stage IIB cervical cancer; stage III cervical cancer; stage IV cervical cancer; stage IVA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — copper(64)TETA-phenyalanyl-tyrosyl(3)-octreotate; Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Copper ATSM (Experimental): pre-therapy pelvic 64Cu-ATSM-PET/CT with Pre- and post- therapy FDG PET/CT
  Interventions: Drug: 64Cu-ATSM; Drug: FDG

INTERVENTIONS:
Drug: 64Cu-ATSM
  Other Names: copper 64; 64Cu Diacetyl-bis(N4-methylthiosemicarbazone)
Drug: FDG
  Other Names: fludeoxyglucose F 18; Fluorodeoxyglucose (18F); 18F-FDG; 18F-fluorodeoxyglucose

SUMMARY:
RATIONALE: Diagnostic procedures, such as 64Cu-labeled diacetyl-bis[N4-methylthiosemicarbazone] (copper Cu 64-ATSM) PET/CT scans, may help doctors predict how patients will respond to treatment.

PURPOSE: This phase II trial is studying how well copper Cu 64-ATSM PET/CT scans work in predicting disease progression in patients undergoing standard of care treatment with cisplatin and radiation therapy (external beam and brachytherapy) per National Comprehensive Cancer Network (NCCN) guidelines for newly-diagnosed stage IB, stage II, stage III, or stage IVA cervical cancer via the Federation of Gynecology and Obstetrics (FIGO) staging systems.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To define the role of pre-therapy ^64Cu-labeled diacetyl-bis(N4-methylthiosemicarbazone) (copper Cu 64-ATSM) in predicting prognosis and determining the behavior of an invasive squamous cell cervical cancer in patients with newly-diagnosed stage IB2-IVA cervical squamous cell carcinoma.
* To determine whether higher copper Cu 64-ATSM uptake is associated with lower progression-free survival of these patients after chemoradiotherapy.

Secondary

* To determine if higher copper Cu 64-ATSM uptake is associated with lower overall survival of these patients.
* To determine if higher copper Cu 64-ATSM uptake is associated with earlier primary cervical tumor recurrence and a higher rate of development of distant metastatic disease in these patients.
* To determine if higher copper Cu 64-ATSM uptake is associated with a lower frequency of complete metabolic response on 2-Deoxy-2-[18F]fluoroglucose (FDG) -PET/CT scan performed 3 months after completion of radiotherapy and chemotherapy.
* To estimate the accuracy of copper Cu 64-ATSM uptake as a predictor of progression-free survival, overall survival, primary tumor recurrence, and future development of distant metastatic disease in these patients.
* To evaluate the performance of copper Cu 64-ATSM uptake as a predictor of lymph node metastasis at study entry.
* To evaluate whether copper Cu 64-ATSM uptake correlates with tumor volume at study entry.
* To examine the relationship between tumor uptake of copper Cu 64-ATSM and other markers of tumor hypoxia, including Vascular endothelial growth factor (VEGF) , Glucose transporter 1 (GLUT1), Carbonic anhydrase IX (CA9/CA IX), and Osteopontin (OPN).
* To compare the predictive ability of pre-therapy copper Cu 64-ATSM-PET to that of post-therapy FDG-PET/CT scan.
* To assess whether pre-therapy FDG-PET/CT findings are predictive of progression-free survival.

OUTLINE: This is a multicenter study.

Patients receive copper Cu 64-ATSM IV and undergo PET/CT scan over 30 minutes 30-40 minutes later. Within 4 weeks after copper Cu 64-ATSM-PET/CT scan, patients begin planned concurrent standard of care chemoradiotherapy comprising 6 weeks of radiotherapy (external beam and brachytherapy)and weekly cisplatin administration per NCCN guidelines. Patients then undergo FDG-PET/CT scan 3 months after completion of chemoradiotherapy.

Tissue samples from previously collected cervical biopsy (obtained for diagnosis) are used for detecting hypoxic markers by immunohistochemistry analysis.

After completion of study intervention, patients are followed for every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary invasive cervical squamous cell carcinoma

  * Newly diagnosed disease
  * Stage IB2 - IVA disease based on FIGO staging system
* Plan to receive standard of care treatment with concurrent cisplatin and radiation therapy (external beam and brachytherapy) per NCCN guidelines

  * Must be scheduled to receive 6 weekly courses of cisplatin
* Meets 1 of the following criteria:

  * Pelvic nodal (or no nodal) disease only by FDG-PET/CT scan within 4 weeks of enrollment
  * Para-aortic nodal metastasis by FDG-PET/CT scan within 4 weeks of enrollment, and patient will undergo radiotherapy to para-aortic nodes
  * FDG-PET/CT scan at baseline if not meeting any of the above criteria
* No stage IVB disease (distant metastases or supraclavicular metastasis) confirmed by FDG-PET/CT scan
* No recurrent invasive carcinoma of the uterine cervix regardless of previous treatment
* No know metastases to lungs, supraclavicular lymph nodes, or other organs outside of the pelvis or abdominal lymph nodes at time of diagnosis

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to lie flat for the duration of the PET/CT scan
* No septicemia or severe infection
* No uncontrolled or poorly controlled diabetes
* No circumstances that would prevent completion of imaging studies or required clinical follow-up
* No other prior or concurrent invasive malignancies, with the exception of non-melanoma skin cancer, within the past 5 years

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior pelvic or abdominal lymphadenectomy
* No prior pelvic radiation therapy
* No previous cancer treatment contraindicates this protocol therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-07-29 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2011-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farrokh Dehdashti, MD, Principal Investigator — Mallinckrodt Institute of Radiology at Washington University Medical Center; David A. Mankoff, MD, PhD, Study Chair — University of Washington
Locations (2):
- United States (2):
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Yes
See NCI data Sharing Policy
Supporting Information: Study Protocol, ICF
Time Frame: July 2009
Access Criteria: Public

REFERENCES:
- See also: National Cancer Institute's Clinical trial database — https://clinicaltrials.gov/ct2/show/NCT00794339

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study funding source changed (from National Cancer Institutes to American College of Radiology Imaging Network foundation) after accrual of 28 individuals
Groups:
- Copper ATSM: pre-therapy pelvic [64Cu][Cu-diacetyl-bis(N(4)-methylthiosemicarbazone)] (64Cu-ATSM) PET/CT exam with Pre- and post- therapy (18)F-fluorodeoxyglucose (FDG) PET/CT exams
Period: Overall Study
Arm/Group | Copper ATSM
Started | 73
Eligible | 69
Evaluable | 59
Completed | 59
Not Completed | 14
Not completed — Withdrawal by Subject | 3
Not completed — Ineligible | 4
Not completed — Tx prior to ATSM | 3
Not completed — ATSM imaging not complete or inadequate | 3
Not completed — Tx not per protocol | 1

BASELINE CHARACTERISTICS:
Population: Eligible evaluable participants
Groups:
- Copper ATSM: pre-therapy pelvic 64Cu-ATSM-PET/CT with Pre- and post- therapy FDG PET/CT
  64Cu-ATSM
  FDG
Arm/Group | Copper ATSM
Number analyzed (Participants) | 59
Age, Continuous [Median (Full Range); unit: years] | 51.2 [25 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 5
  White | 39
  More than one race | 0
  Unknown or Not Reported | 11
FIGO stage [Count of Participants; unit: Participants] — Fédération Internationale de Gynécologie et d'Obstétrique (FIGO) stage is divided into 5 primary stages(and subtypes A &B within each category), with stage 5 being the most severe.
  stage 0: carcinoma in situ stage I: confined to the organ of origin stage II: invasion of surrounding organs or tissue stage III: spread to distant nodes or tissue within the pelvis stage IV: distant metastasis(es)
  Participants
    IB2 | 15
    IIA | 5
    IIB | 21
    III | 1
    IIIA | 2
    IIIB | 12
    IVA | 3

OUTCOME MEASURES:

1. Primary Outcome: Relationship Between Copper Cu 64-ATSM Uptake in the Primary Tumor and Progression-free Survival 3 Years After Chemoradiotherapy
Description: Progression-free survival (PFS) evaluated every 3 months for first 2 years and every 6 months during year 3 to determine PFS at 3years.
  Cu64-ATSM Uptake measured within 14 days of baseline Uptake is a measure of activity within a tumor
  1. the maximum standardized uptake value (SUVmax = tracer uptake in ROI / (injected activity / patient weight))
  2. Tumor-to-Muscle uptake ratio (T/M, An FDG-PET/CT-guided circular region of interest of 1.0-1.5 cm in diameter is drawn around the most intense region of the primary tumor to calculate the maximum uptake within the region. In addition, regions of interest are drawn on bilateral gluteal muscle groups on at least 3 slices, and the mean uptake is calculated. The T/M is the ratio of these measurements.)
Time Frame: every 3 months for first 2 years and every 6 months during year 3, up to 3 years
Population: As a fully paired analysis, all participants were evaluated in each group. 21 participants progressed by year 3 and 38 participants were progression free at year 3.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- 64 CU-ATSM SUVmax @ Baseline: The maximum standardized uptake value (SUVmax) is the Cu64-ATSM Uptake measured within 14 days of baseline is defined as SUVmax = tracer uptake in ROI / (injected activity / patient weight))
- 64 CU-ATSM T/M Ratio @ Baseline: Cu64-ATSM uptake measured using the Tumor-to-Muscle uptake ratio within 14 days of baseline The tumor uptake is measured by selecting an FDG-PET/CT-guided circular region of interest of 1.0-1.5 cm in diameter around the most intense region of the primary tumor to calculate the maximum uptake within the region.
  The Muscle uptake is measured by selecting regions of interest on bilateral gluteal muscle groups on at least 3 slices, and calculating the mean uptake.
  The T/M uptake is the ratio of these 2 measurements.
Arm/Group | 64 CU-ATSM SUVmax @ Baseline | 64 CU-ATSM T/M Ratio @ Baseline
Number analyzed (Participants) | 59 | 59
ratio
  Progression within 3 years: number analyzed (Participants) | 21 | 21
  Progression within 3 years | 4.4 (1.3) | 8.2 (4.1)
  No progression within 3 years: number analyzed (Participants) | 38 | 38
  No progression within 3 years | 4.2 (1.3) | 8.0 (3.1)

2. Secondary Outcome: Copper Cu 64-ATSM T/M Uptake and Overall Survival
Description: To determine if higher 64Cu-ATSM uptake on PET/CT is associated with lower Overall survival (OS) T/M Uptake measured within 14 days of baseline;
  Overall survival (OS) is measured every 3 months for first 2 years and every 6 months during year 3,until time of death or 3 years from baseline.
Time Frame: every 3 months for first 2 years and every 6 months during year 3, up to 3 years
Population: Participants were divided into two groups by whether their T/M Ratio fell at or above vs. below the observed median of 7.3.
Measure: Median (Full Range); unit: days
Groups:
- T/M Below Median: Tumor-to-muscle ratio (T/M) below the observed median value of 7.3
- T/M at or Above Median: Tumor-to-muscle ratio (T/M) at or above the observed median value of 7.3
Arm/Group | T/M Below Median | T/M at or Above Median
Number analyzed (Participants) | 28 | 31
days | 773.5 [46 to 1378] | 786.0 [14 to 1196]
Statistical Analysis 1: Comparison: T/M Below Median vs T/M at or Above Median; Participants were divided into two groups by whether their T/M Ratio fell at or above vs. below the observed median of 7.3 and the the median survival was compared between the 2 groups; Test type: Equivalence — equivalence margin=0; p = 0.4883, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Relationship Between Copper Cu 64-ATSM Uptake and Complete Metabolic Response
Description: Complete metabolic response determined by FDG PET/CT performed 3 months after completion of chemoradiation By definition, metabolic response (as defined by NCI Concept ID: C3897320. https://www.ncbi.nlm.nih.gov/medgen/856914) is "the disappearance of metabolic tumor activity in target and non-target lesions, marked by a decrease in tumor standardized uptake value to the level of surrounding normal tissue (tumor uptake/normal uptake = ~1)"
Time Frame: 3 months after completion of chemoradiation
Population: 52 observations were used for this analysis. 7 participants did not have FDG PET data available for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: All eligible participants with evaluable pre-therapy pelvic 64Cu-ATSM-PET/CT within 14 days of baseline and with Pre- and post- therapy FDG PET/CT
Arm/Group | Eligible Participants
Number analyzed (Participants) | 52
Participants
  Complete metabolic response | 23
  Partial response or progressive disease | 29
Statistical Analysis 1: Comparison: Eligible Participants; Logistic Regression Modeling Complete Metabolic Response by T/M Ratio; Test type: Equivalence — no equivalence margin; p = 0.1924, Regression, Logistic; Slope = -0.1235, Standard Error of Mean 1.6988

4. Secondary Outcome: Primary Tumor Recurrence
Description: To determine if higher 64Cu ATSM uptake is associated with earlier primary cervical tumor recurrence images were taken every 3 months for first 2 years and every 6 months during year 3, up to 3 years and evaluated for primary cervical tumor recurrence
Time Frame: every 3 months for first 2 years and every 6 months during year 3, up to 3 years
Population: Two participants were off study before the follow up period began (one death and one withdrawal) and were not assessed for disease status - thus only 57 of the 59 participants were evaluated for this outcome.
Measure: Median (Full Range); unit: days
Arm/Group | T/M Below Median | T/M at or Above Median
Number analyzed (Participants) | 28 | 29
days | 773.5 [46 to 1378] | 797.0 [252 to 1196]
Statistical Analysis 1: Comparison: T/M Below Median vs T/M at or Above Median; Participants were divided into two groups: those at or above the median for T/M Ratio (7.3) vs. those below, and the time to primary tumor recurrence was compared between the 2 goups; Test type: Equivalence — equivalence margin = 0; p = 0.3090, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Lymph Node Metastasis at Baseline
Description: Lymph nodes were evaluated at 5 locations: Pelvic, Common Iliac, Para Aortic, Mediastinal, and Supraclavicular
  This outcome looks at the Association of Ratio of Tissue to Muscle (T/M) uptake with Lymph Node Metastases at Baseline
Time Frame: Two weeks
Population: one patient's scan could not evaluated for any lymph nodes, and three others could be evaluated only for pelvic lymph nodes.
Measure: Count of Participants; unit: Participants
Arm/Group | Eligible Participants
Number analyzed (Participants) | 58
Participants
  Pelvic: Positive Nodes | 31
  Pelvic: Negative Nodes | 27
  Common Iliac: number analyzed (Participants) | 55
  Common Iliac: Positive Nodes | 14
  Common Iliac: Negative Nodes | 41
  Para Aortic: number analyzed (Participants) | 55
  Para Aortic: Positive Nodes | 7
  Para Aortic: Negative Nodes | 48
  Mediastinal: number analyzed (Participants) | 55
  Mediastinal: Positive Nodes | 0
  Mediastinal: Negative Nodes | 55
  Supraclavicular: number analyzed (Participants) | 55
  Supraclavicular: Positive Nodes | 0
  Supraclavicular: Negative Nodes | 55
Statistical Analysis 1: Comparison: Eligible Participants; Logistic Regression Evaluating Tissue to Muscle (T/M) uptake ratio as a Predictor of PELVIC Lymph Node Metastases at Baseline; Test type: Equivalence — equivalence margin=0; p = 0.5291, Regression, Logistic
Statistical Analysis 2: Comparison: Eligible Participants; Logistic Regression Evaluating Tissue to Muscle (T/M) uptake Ratio as a Predictor of COMMON ILIAC Lymph Node Metastases at Baseline; Test type: Equivalence — equivalence margin=0; p = 0.9684, Regression, Logistic
Statistical Analysis 3: Comparison: Eligible Participants; Logistic Regression Evaluating Tissue to Muscle (T/M) uptake Ratio as a Predictor of Para Aortic Lymph Node Metastases at Baseline; Test type: Equivalence — equivalence margin=0; p = 0.7327, Regression, Logistic

6. Secondary Outcome: Relationship of Copper Cu 64-ATSM Uptake T/M Ratio and Carbonic Anhydrase IX (CA-IX) Percentage of Tumor Cells Staining Score as a Marker of Tumor Hypoxia
Description: The Ratio of Tissue to Muscle (T/M) agent uptake measured at baseline was used as a predictor of Hypoxia Tumor Hypoxia was assessed with Carbonic anhydrase IX (CA-IX) markers using the
  Percentage of Tumor Cells Staining Score:
  0=<1% tumor cells; 1=1 33% tumor cells; 2=34 66% tumor cells; and 3=>66% tumor cells.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- 0=<1% Tumor Cells: T/M ratio for subjects with Hypoxia categorized as 0=<1% tumor cells using the Percentage of Tumor Cells Staining Score.
- 1-33% Tumor Cells: T/M ratio for subjects with Hypoxia categorized as 1-33% tumor cells using the Percentage of Tumor Cells Staining Score.
- 34-66% Tumor Cells: T/M ratio for subjects with Hypoxia categorized as 34-66% tumor cells using the Percentage of Tumor Cells Staining Score.
- >66% Tumor Cells: T/M ratio for subjects with Hypoxia categorized as >66% tumor cells using the Percentage of Tumor Cells Staining Score.
Arm/Group | 0=<1% Tumor Cells | 1-33% Tumor Cells | 34-66% Tumor Cells | >66% Tumor Cells
Number analyzed (Participants) | 16 | 17 | 13 | 2
ratio | 7.58 (2.87) | 7.57 (3.17) | 9.40 (5.26) | 7.35 (1.20)

7. Secondary Outcome: Relationship of Copper Cu 64-ATSM Uptake T/M Ratio and CA-IX Staining Intensity Score: as a Marker of Tumor Hypoxia
Description: The Ratio of Tissue to Muscle (T/M) agent uptake measured at baseline was used as a predictor of Hypoxia Tumor Hypoxia was assessed with CA-IX markers using the
  Staining Intensity Score:
  0=No staining; 1=Weak staining; and 2=Moderate to strong staining.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- No Staining: T/M ratio for subjects with Hypoxia categorized as "No staining" using the Staining Intensity Score
- Weak Staining: T/M ratio for subjects with Hypoxia categorized as "Weak staining" using the Staining Intensity Score
- Moderate to Strong Staining: T/M ratio for subjects with Hypoxia categorized as "Moderate to strong staining" using the Staining Intensity Score
Arm/Group | No Staining | Weak Staining | Moderate to Strong Staining
Number analyzed (Participants) | 16 | 11 | 21
ratio | 7.58 (2.87) | 6.20 (2.56) | 9.40 (4.37)

8. Secondary Outcome: Relationship of Copper Cu 64-ATSM Uptake T/M Ratio and CA-IX Composite Score as a Marker of Tumor Hypoxia
Description: The Ratio of Tissue to Muscle (T/M) agent uptake measured at baseline was used as a predictor of Hypoxia Tumor Hypoxia was assessed with CA-IX markers using the
  Composite Score (range 0-6):
  Computed by using the coded values of Percentage of Tumor Cells Staining Score (0-3) multiplied by the coded value of Staining Intensity Score (0-2).
Time Frame: Baseline
Population: No cases had a composite score of 5
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Composite Score: 0: T/M ratio for subjects with Hypoxia composite score of 0
- Composite Score: 1: T/M ratio for subjects with Hypoxia composite score of 1
- Composite Score: 2: T/M ratio for subjects with Hypoxia composite score of 2
- Composite Score: 3: T/M ratio for subjects with Hypoxia composite score of 3
- Composite Score: 4: T/M ratio for subjects with Hypoxia composite score of 4
- Composite Score: 6: T/M ratio for subjects with Hypoxia composite score of 6
Arm/Group | Composite Score: 0 | Composite Score: 1 | Composite Score: 2 | Composite Score: 3 | Composite Score: 4 | Composite Score: 6
Number analyzed (Participants) | 16 | 6 | 15 | 1 | 9 | 1
ratio | 7.58 (2.87) | 5.82 (1.99) | 8.04 (3.44) | 6.50 (NA) — SD cannot be computed with 1 observation | 10.60 (5.54) | 8.20 (NA) — SD cannot be computed with 1 observation

9. Secondary Outcome: Relationship of Copper Cu 64-ATSM Uptake T/M Ratio and VEGF Percentage of Tumor Cells Staining Score as a Marker of Tumor Hypoxia
Description: The Ratio of Tissue to Muscle (T/M) agent uptake measured at baseline was used as a predictor of Hypoxia Tumor Hypoxia was assessed with VEGF markers using the
  Percentage of Tumor Cells Staining Score:
  0=<1% tumor cells; 1=1 33% tumor cells; 2=34 66% tumor cells; and 3=>66% tumor cells.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 0=<1% Tumor Cells | 1-33% Tumor Cells | 34-66% Tumor Cells | >66% Tumor Cells
Number analyzed (Participants) | 11 | 4 | 19 | 14
ratio | 6.98 (2.54) | 7.57 (4.57) | 8.51 (3.65) | 8.44 (4.50)

10. Secondary Outcome: Relationship of Copper Cu 64-ATSM Uptake T/M Ratio and Vascular Endothelial Growth Factor (VEGF) Staining Intensity Score: as a Marker of Tumor Hypoxia
Description: The Ratio of Tissue to Muscle (T/M) agent uptake measured at baseline was used as a predictor of Hypoxia Tumor Hypoxia was assessed with Vascular endothelial growth factor (VEGF) markers using the
  Staining Intensity Score:
  0=No staining; 1=Weak staining; and 2=Moderate to strong staining.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | No Staining | Weak Staining | Moderate to Strong Staining
Number analyzed (Participants) | 11 | 25 | 12
ratio | 6.98 (2.54) | 7.50 (3.17) | 10.22 (4.93)

11. Secondary Outcome: Relationship of Copper Cu 64-ATSM Uptake T/M Ratio and Vascular Endothelial Growth Factor (VEGF) Composite Score as a Marker of Tumor Hypoxia
Description: The Ratio of Tissue to Muscle (T/M) agent uptake measured at baseline was used as a predictor of Hypoxia Tumor Hypoxia was assessed with Vascular endothelial growth factor (VEGF) markers using the
  Composite Score (range 0-6):
  Computed by using the coded values of Percentage of Tumor Cells Staining Score (0-3) multiplied by the coded value of Staining Intensity Score (0-2).
Time Frame: Baseline
Population: No cases had a composite score of 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Composite Score: 0 | Composite Score: 1 | Composite Score: 2 | Composite Score: 3 | Composite Score: 4 | Composite Score: 6
Number analyzed (Participants) | 11 | 2 | 16 | 9 | 5 | 5
ratio | 6.98 (2.54) | 4.44 (1.22) | 8.79 (3.67) | 6.59 (1.83) | 8.48 (4.11) | 11.76 (6.13)

12. Secondary Outcome: Relationship of Copper Cu 64-ATSM Uptake T/M Ratio and Glucose Transporter 1 (GLUT1) Percentage of Tumor Cells Staining Score as a Marker of Tumor Hypoxia
Description: The Ratio of Tissue to Muscle (T/M) agent uptake measured at baseline was used as a predictor of Hypoxia Tumor Hypoxia was assessed with Glucose transporter 1 (GLUT1) markers using the
  Percentage of Tumor Cells Staining Score:
  0=<1% tumor cells; 1=1 33% tumor cells; 2=34 66% tumor cells; and 3=>66% tumor cells.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | 0=<1% Tumor Cells | 1-33% Tumor Cells | 34-66% Tumor Cells | >66% Tumor Cells
Number analyzed (Participants) | 2 | 5 | 23 | 18
ratio | 9.70 (0.42) | 6.01 (1.08) | 8.83 (4.22) | 7.46 (3.49)

13. Secondary Outcome: Relationship of Copper Cu 64-ATSM Uptake T/M Ratio and Glucose Transporter 1 (GLUT1) Staining Intensity Score: as a Marker of Tumor Hypoxia
Description: The Ratio of Tissue to Muscle (T/M) agent uptake measured at baseline was used as a predictor of Hypoxia Tumor Hypoxia was assessed with GLUT-1 markers using the
  Staining Intensity Score:
  0=No staining; 1=Weak staining; and 2=Moderate to strong staining.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | No Staining | Weak Staining | Moderate to Strong Staining
Number analyzed (Participants) | 2 | 6 | 40
ratio | 9.70 (0.42) | 7.15 (1.47) | 8.11 (4.01)

14. Secondary Outcome: Relationship of Copper Cu 64-ATSM Uptake T/M Ratio and Glucose Transporter 1 (GLUT1) Composite Score as a Marker of Tumor Hypoxia
Description: The Ratio of Tissue to Muscle (T/M) agent uptake measured at baseline was used as a predictor of Hypoxia Tumor Hypoxia was assessed with Glucose transporter 1 (GLUT1) markers using the
  Composite Score (range 0-6):
  Computed by using the coded values of Percentage of Tumor Cells Staining Score (0-3) multiplied by the coded value of Staining Intensity Score (0-2).
Time Frame: Baseline
Population: No cases had a composite score of 5
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Composite Score: 0 | Composite Score: 1 | Composite Score: 2 | Composite Score: 3 | Composite Score: 4 | Composite Score: 6
Number analyzed (Participants) | 2 | 2 | 6 | 1 | 20 | 17
ratio | 9.70 (0.42) | 6.55 (0.07) | 6.89 (1.84) | 5.40 (NA) — SD cannot be computed with 1 observation | 8.93 (4.50) | 7.58 (3.56)

15. Secondary Outcome: Relationship Between Copper Cu 64-ATSM Uptake and Development of Distant Metastasis
Description: Existence of distant metastasis was evaluated every 3 months for first 2 years and every 6 months during year 3 Copper Cu 64-ATSM Uptake (T/M) measured within 14 days of baseline;
Time Frame: every 3 months for first 2 years and every 6 months during year 3, up to 3 years
Population: Participants were divided into two groups by whether their T/M Ratio fell at or above vs. below the observed median of 7.3 and the median time (days) was calculated for the development of new distant metastases.
Measure: Median (Full Range); unit: days
Arm/Group | T/M Below Median | T/M at or Above Median
Number analyzed (Participants) | 28 | 31
days | 725.5 [46 to 1378] | 786.0 [138 to 1196]
Statistical Analysis 1: Comparison: T/M Below Median vs T/M at or Above Median; Participants were divided into two groups by whether their T/M Ratio fell at or above vs. below the observed median of 7.3 and the time to observe new distant metastases was compared between the groups; Test type: Equivalence — equivalence margin=0; p = .4981, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: within 24 hours of 64Cu-ATSM administration
Description: Any death or AE occurring at any time after a participant has discontinued or terminated study participation that might be reasonably related to the 64Cu-ATSM-PET/CT trial was to be reported.
Arm/Group | Copper ATSM
All-Cause Mortality (participants affected / at risk) | 0/59
Serious Adverse Events (participants affected / at risk) | 0/59
Other Adverse Events (participants affected / at risk) | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No